CLINICAL TRIAL: NCT02557516
Title: Open Label 1b/2a Trial of a Combination of IPH2201 and Ibrutinib in Patients With Relapsed, Refractory or Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: Combination Study of IPH2201 (Monalizumab) With Ibrutinib in Relapsed, Refractory or Previously Untreated CLL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IPH2201-202
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — monalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase 1 Level 1 - 1 mg/kg (Experimental): In phase 1, Monalizumab given at the first dose level of 1 mg/kg.
  Interventions: Drug: monalizumab
- Phase 1 Level 2 - 2 mg/kg (Experimental): In phase 1, Monalizumab given at the second dose level of 2 mg/kg.
  Interventions: Drug: monalizumab
- Phase 1 Level 3 - 4 mg/kg (Experimental): In phase 1, Monalizumab given at the third dose level of 4 mg/kg.
  Interventions: Drug: monalizumab
- Phase 2 RP2D - 2 mg/kg (Experimental): In phase 2, Monalizumab given at the Recommended Phase 2 Dose (RP2D) of 2 mg/kg, selected by a safety committee.
  Interventions: Drug: monalizumab

INTERVENTIONS:
Drug: monalizumab — During phase 1, patients received monalizumab, IV, at the dose of 1, 2 or 4mg/kg, as a single agent during 4 weeks and thereafter combined with ibrutinib 420 mg, orally, once daily, during 52 weeks.
  During phase 2, patients received monalizumab, IV, at the dose recommended upon completion of phase 1, combined with ibrutinib 420 mg orally, once daily, from the first cycle, during 52 weeks. In both parts of the trial, the first 4 administrations of monalizumab (from week 0 to week 6) occured every 2 weeks. From the 5th administration monalizumab was administered every 4 weeks.
  Other Names: Anti-NKG2A; IPH2201

SUMMARY:
Combination study of monalizumab (IPH2201) with Ibrutinib in relapsed, refractory or previously untreated Chronic Lymphocytic Leukemia (CLL) patients in 2 parts :

* phase 1 : a 3+3 design to assess the Maximum Tolerated Dose (MTD)
* phase 2: to evaluate the anti-leukemic activity of the combination

DETAILED DESCRIPTION:
This trial was designated to test the hypothesis that the combination of ibrutinib and IPH2201 will result in a substantial complete response (CR) rate, especially CR without minimal residual disease (MRD), as this has been shown to be associated with long-term clinical benefit.

Up to 45 patients were planned to be enrolled. During the phase 1 part a 3+3 dose escalation design was employed. Four doses were planned to be assessed if the Maximum Tolerated Dose (MTD) was not previously reached: 1, 2, 4 and 10 mg/kg.

During phase 2 part, patients received monalizumab in combination with ibrutinib; monalizumab was given at the dose recommended upon completion of the phase I portion.

The primary objective of the phase 1 was to assess the safety of monalizumab given intravenously as a single agent and in combination with ibrutinib in patients with relapsed, refractory or previously untreated Chronic Lymphocytic Leukemia.

The primary objective of the phase 2 was to evaluate the anti-leukemic activity of the combination of monalizumab and ibrutinib in patients with relapsed, refractory or previously untreated Chronic Lymphocytic Leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Chronic Lymphocytic Leukemia (CLL)
* Relapsed, refractory or previously untreated CLL
* CLL requiring treatment; patients must be eligible for ibrutinib therapy
* Age > = 18 years
* Eastern Cooperative Oncology Group performance status of 0-2
* Life expectancy > = 3 months
* Adequate liver and renal function
* Negative serum pregnancy test within 72 hours before starting study treatment in women with childbearing potential. Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of the study participation
* Ability to understand a written informed and consent document
* Signed informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* Patients who have previously received ibrutinib or another inhibitor of Bruton's tyrosine kinase (BTK)
* History of allergic reactions attributed to compounds or similar chemical or biological composition to ibrutinib
* Central nervous system involvement of the CLL
* Abnormal hematological function which is not due to bone marrow failure related to the CLL
* Patients requiring a treatment by oral vitamin K antagonists
* Serious uncontrolled medical disorder
* Medical condition or organ system dysfunction which, in the investigator opinion, could interfere with absorption or metabolism of ibrutinib
* Moderate or severe hepatic impairment
* Active auto-immune disease
* Abnormal cardiac status
* Pregnant women are excluded from study
* Current active infectious disease
* History of another malignancy within 3 years
* History of allogeneic stem cell or solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2019-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry A Rogers, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was anticipated that up to 24 patients (3 to 6 patients; 4 dose levels) would be enrolled in Phase 1 part of the study and up to 24 patients in the Phase 2 part with a total of up to 45 patients in the trial.
  A total of 22 patients were actually enrolled in the study: 13 patients in the Phase 1 part and 9 patients in the Phase 2 part.
Pre-assignment Details: The first part of the study had a 3+3 design. Four dose levels of monalizumab were planned: 1 mg/kg, 2 mg/kg, 4 mg/kg and 10 mg/kg. Dose-escalation decisions were made by a Safety Committee.The dose of monalizumab for all patients in phase 2 of the study (2 mg/kg) was also chosen by the Safety Committee based on phase 1 data.
Groups:
- Phase 1 Level 1 - 1 mg/kg: During phase 1, patients received monalizumab, IV, at the dose of 1mg/kg, as a single agent during 4 weeks and thereafter combined with ibrutinib 420 mg, orally, once daily, during 52 weeks.
  The first 4 administrations of monalizumab occured every 2 weeks. From the 5th administration monalizumab was administered every 4 weeks.
- Phase 1 Level 2 - 2 mg/kg: During phase 1, patients received monalizumab, IV, at the dose of 2 mg/kg, as a single agent during 4 weeks and thereafter combined with ibrutinib 420 mg, orally, once daily, during 52 weeks.
  The first 4 administrations of monalizumab occured every 2 weeks. From the 5th administration monalizumab was administered every 4 weeks.
- Phase 1 Level 3 - 4 mg/kg: During phase 1, patients received monalizumab, IV, at the dose of 4 mg/kg, as a single agent during 4 weeks and thereafter combined with ibrutinib 420 mg, orally, once daily, during 52 weeks.
  The first 4 administrations of monalizumab occured every 2 weeks. From the 5th administration IPH2201 was administered every 4 weeks.
- Phase 2 RP2D - 2 mg/kg: During phase 2, patients received monalizumab, IV, at the dose recommended upon completion of phase 1 part (2 mg/kg), combined with ibrutinib 420 mg orally, once daily, from the first administration and during 52 weeks.
  The first 4 administrations of monalizumab occured every 2 weeks. From the 5th administration monalizumab was administered every 4 weeks.
Period: Overall Study
Arm/Group | Phase 1 Level 1 - 1 mg/kg | Phase 1 Level 2 - 2 mg/kg | Phase 1 Level 3 - 4 mg/kg | Phase 2 RP2D - 2 mg/kg
Started | 3 | 6 | 4 | 9
Completed | 2 | 1 | 0 | 0
Not Completed | 1 | 5 | 4 | 9
Not completed — Adverse Event | 1 | 0 | 2 | 1
Not completed — Disease progression | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0
Not completed — Sponsor decision | 0 | 1 | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Phase 1 Level 1 - 1 mg/kg: During phase 1, patients received monalizumab, IV, at the dose of 1 mg/kg, as a single agent during 4 weeks and thereafter combined with ibrutinib 420 mg, orally, once daily, during 52 weeks.
  In both parts of the trial, the first 4 administrations of monalizumab occured every 2 weeks. From the 5th administration monalizumab was administered every 4 weeks.
- Phase 1 Level 2 - 2 mg/kg: During phase 1, patients received monalizumab, IV, at the dose of 2 mg/kg, as a single agent during 4 weeks and thereafter combined with ibrutinib 420 mg, orally, once daily, during 52 weeks.
  In both parts of the trial, the first 4 administrations of monalizumab occured every 2 weeks. From the 5th administration monalizumab was administered every 4 weeks.
- Phase 1 Level 3 - 4 mg/kg: During phase 1, patients received monalizumab, IV, at the dose of 4 mg/kg, as a single agent during 4 weeks and thereafter combined with ibrutinib 420 mg, orally, once daily, during 52 weeks.
  In both parts of the trial, the first 4 administrations of monalizumab occured every 2 weeks. From the 5th administration monalizumab was administered every 4 weeks.
- Phase 2 RP2D - 2 mg/kg: During phase 2, patients received monalizumab, IV, at the dose recommended upon completion of phase 1 part, combined with ibrutinib 420 mg orally, once daily, from the first cycle and during 52 weeks.
  In both parts of the trial, the first 4 administrations of monalizumab occured every 2 weeks. From the 5th administration monalizumab was administered every 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Level 1 - 1 mg/kg | Phase 1 Level 2 - 2 mg/kg | Phase 1 Level 3 - 4 mg/kg | Phase 2 RP2D - 2 mg/kg | Total
Number analyzed (Participants) | 3 | 6 | 4 | 9 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (11.15) | 65.8 (7.14) | 69.5 (10.08) | 69.4 (6.33) | 67.1 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3 | 2 | 8
  Male | 3 | 3 | 1 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 4 | 9 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 3 | 6 | 4 | 7 | 20
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 4 | 9 | 22
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group performance status scale 0 Fully active, able to carry out all normal activity without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out light work.
  2. Ambulatory and capable of all self-care but unable to carry out any work. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care, confined to bed or chair more than 50 % of waking hours.
  4. Completely disabled. Cannot carry out any self-care. Totally confined to bed or chair.
  5. Dead.
  Participants
    ECOG 0 | 3 | 2 | 0 | 7 | 12
    ECOG 1 | 0 | 4 | 4 | 2 | 10
RAI Stage [Count of Participants; unit: Participants] — The RAI staging divides CLL into 5 stages:
  stage 0, bone marrow and blood lymphocytosis only; stage I, lymphocytosis with enlarged nodes; stage II, lymphocytosis with enlarged spleen or liver or both; stage III, lymphocytosis with anemia; and stage IV:lymphocytosis with thrombocytopenia.
  Stage 0 is low-risk, stages I and II are intermediate-risk, stages III and IV are high-risk.
  Participants
    Stage I | 0 | 0 | 0 | 3 | 3
    Stage II | 2 | 1 | 0 | 0 | 3
    Stage III | 0 | 1 | 1 | 0 | 2
    Stage IV | 1 | 4 | 3 | 6 | 14
Disease Status at Screening [Count of Participants; unit: Participants]
  Previously Untreated CLL | 0 | 1 | 0 | 6 | 7
  Refractory CLL | 0 | 1 | 1 | 0 | 2
  Relapse CLL | 3 | 4 | 3 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities
Description: Number of dose-limiting toxicities, measured during the phase 1, dose escalation, part of the study.
Time Frame: 8 weeks
Population: During phase 1 part of the study (dose escalation) the total number of patients evaluated for safety parameters is 13; 3 patients received at least one dose of monalizumab 1 mg/kg, 6 patients received 2 mg/kg , and 4 patients received 4 mg/kg.
Measure: Number; unit: Dose Limiting Toxicy
Groups:
- Phase 1 Level 1 - 1 mg/kg: Phase 1 (dose escalation) evaluating dose level 1 (1 mg/kg) of monalizumab alone during 4 weeks then in combination with ibrutinib during 52 weeks.
- Phase 1 Level 2 - 2 mg/kg: Phase 1 (dose escalation) evaluating dose level 2 of monalizumab (2 mg/kg) of monalizumab alone during 4 weeks then in combination with ibrutinib during 52 weeks.
- Phase 1 Level 3 - 4 mg/kg: Phase 1 (dose escalation) evaluating dose level 3 (4 mg/kg) of monalizumab alone during 4 weeks then in combination with ibrutinib during 52 weeks.
Arm/Group | Phase 1 Level 1 - 1 mg/kg | Phase 1 Level 2 - 2 mg/kg | Phase 1 Level 3 - 4 mg/kg
Number analyzed (Participants) | 3 | 6 | 4
Dose Limiting Toxicy | 0 | 1 | 2

2. Primary Outcome: Rate of Complete Response (CR)
Description: The rate of complete response (CR) was evaluated using the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) grading scale and confirmed by a bone marrow biopsy. Per International Workshop on Chronic Lymphocytic Leukemia (IWCLL), Complete Response (CR) is defined as lymphocytes <4x109/l, absence of lymphadenopathy, hepatomegaly and splenomegaly at CT scan, no constitutional symptoms, no cytopenia, normocellular bone marrow. Partial Response (PR) is a reduction > 50% in lymphocytes, lymphadenopathy, spleen or liver, no cytopenia. PD if appearance of any new lesion, or increase in lymphocytes > 50%, or occurrence of cytopenia attributable to CLL.
Time Frame: CR assessed 52 weeks after the beginning of combination treatment
Population: Efficacy population: 21 patients who received at least one dose of monalizumab. According to the protocol, patients who discontinued treatment due to disease progression before the end of 8 weeks were replaced. Of note,1 patient (grade 3 hemolytic anemia due to disease progression at W4) was replaced and was then excluded from efficacy population.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Level 1 - 1 mg/kg: During phase 1b, patients received monalizumab, IV, at the dose of 1mg/kg, as a single agent during 4 weeks and thereafter combined with ibrutinib 420 mg, orally, once daily, during 52 weeks.
  In both parts of the trial, the first 4 administrations of IPH2201 occured every 2 weeks. From the 5th administration monalizumab was administered every 4 weeks.
- Phase 1 Level 2 - 2 mg/kg: During phase 1b, patients received monalizumab, IV, at the dose of 2 mg/kg, as a single agent during 4 weeks and thereafter combined with ibrutinib 420 mg, orally, once daily, during 52 weeks.
  In both parts of the trial, the first 4 administrations of IPH2201 occured every 2 weeks. From the 5th administration monalizumab was administered every 4 weeks.
- Phase 1 Level 3 - 4 mg/kg: During phase 1b, patients received monalizumab, IV, at the dose of 4 mg/kg, as a single agent during 4 weeks and thereafter combined with ibrutinib 420 mg, orally, once daily, during 52 weeks.
  In both parts of the trial, the first 4 administrations of IPH2201 occured every 2 weeks. From the 5th administration monalizumab was administered every 4 weeks.
- Phase 2 RP2D - 2 mg/kg: During phase 2a, patients received monalizumab, IV, at the dose recommended upon completion of phase 1b part, combined with ibrutinib 420 mg orally, once daily, from the first cycle and during 52 weeks.
  In both parts of the trial, the first 4 administrations of IPH2201 occured every 2 weeks. From the 5th administration monalizumab was administered every 4 weeks
Arm/Group | Phase 1 Level 1 - 1 mg/kg | Phase 1 Level 2 - 2 mg/kg | Phase 1 Level 3 - 4 mg/kg | Phase 2 RP2D - 2 mg/kg
Number analyzed (Participants) | 3 | 6 | 3 | 9
Participants | 1 | 1 | 0 | 0

3. Secondary Outcome: Best Overall Response / Remission Rates
Description: Measure of best overall response at any time during the study. cCR: confirmed complete response/remission; uCR: unconfirmed complete response / remission; PR: partial response/remission; SD: stable disease; PD: progressive disease.
  Per International Workshop on Chronic Lymphocytic Leukemia (IWCLL), Complete Response (CR) is defined as lymphocytes <4x109/l, absence of lymphadenopathy, hepatomegaly and splenomegaly at CT scan, no constitutional symptoms, no cytopenia, normocellular bone marrow. Partial Response (PR) is a reduction > 50% in lymphocytes, lymphadenopathy, spleen or liver, no cytopenia. PD if appearance of any new lesion, or increase in lymphocytes > 50%, or occurrence of cytopenia attributable to CLL.
  In order to have a confirmed CR (cCR), the CR must be confirmed by a scan and a bone marrow assessment assessed at least 2 months after the first occurrence of CR. Otherwise it would be an unconfirmed CR (uCR).
Time Frame: From beginning of study drug treatment to the end of study (up to 24 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Level 3 - 4 mg/kg: During phase 1, patients receive monalizumab, IV, at the dose of 4 mg/kg, as a single agent during 4 weeks and thereafter combined with ibrutinib 420 mg, orally, once daily, during 52 weeks.
  In both parts of the trial, the first 4 administrations of monalizumab occured every 2 weeks. From the 5th administration monalizumab was administered every 4 weeks.
- Phase 2 RP2D - 2 mg/kg: During phase a, patients received monalizumab, IV, at the dose recommended upon completion of phase 1, combined with ibrutinib 420 mg orally, once daily, from the first cycle and during 52 weeks.
  In both parts of the trial, the first 4 administrations of monalizumab occured every 2 weeks. From the 5th administration monalizumab was administered every 4 weeks.
Arm/Group | Phase 1 Level 1 - 1 mg/kg | Phase 1 Level 2 - 2 mg/kg | Phase 1 Level 3 - 4 mg/kg | Phase 2 RP2D - 2 mg/kg
Number analyzed (Participants) | 3 | 6 | 3 | 9
Participants
  cCR | 1 | 1 | 0 | 0
  uCR | 0 | 1 | 0 | 0
  PR | 2 | 3 | 2 | 6
  SD | 0 | 1 | 1 | 3
  PD | 0 | 0 | 0 | 0

4. Secondary Outcome: Duration of Remission
Description: The duration of remission (DOR) is defined as the time from the date of first evaluation of the remission (cCR, uCR or PR) to the first documentation of progressive disease, relapsed disease or death. In case an assessment of progressive / relapsed disease or death does not exist, the DOR was censored at the time of the last disease assessment date. The DOR was calculated only for the patients with a remission that was assessed at 52 weeks.
Time Frame: Up to 24 months
Population: 21 patients evaluated for efficacy. 1 patient treated at 4 mg/kg was withdrawn due to grade 3 hemolytic anemia attribuated to disease progression at W4 and considered as not evaluable for efficacy. Due to the small size of the trial no subgroup analyses have been conducted.
Measure: Median (95% Confidence Interval); unit: Month
Groups:
- Efficacy Population: The efficacy population included all patients who have received at least one dose of monalizumab.
  According to the protocol, patients who discontinued from monalizumab treatment due to disease progression before the end of 8 weeks of treatment were replaced. As one patient was withdrawn due to grade 3 hemolytic anemia attribuated to disease progressions at W4, 21 patients were included in the efficacy population.
Arm/Group | Efficacy Population
Number analyzed (Participants) | 21
Month | NA [NA to NA] — A median DOR could not be estimated at the time of data cut-off.

5. Secondary Outcome: Progression Free Survival
Description: The Progression Free Survival (PFS) is defined as the time from first dose administration until the occurrence of progressive disease, relapsed disease or death from any cause. Patients without an event at the time of the analyse were censored at his or her last disease assessment date. Patients with no post-Baseline assessment were censored at the day of the first dose administration.
Time Frame: Up to 24 months
Population: All 22 enrolled patients were included in the ITT / Safety population
Measure: Median (95% Confidence Interval); unit: Month
Groups:
- ITT / Safety Population: The Intent-To-Treat / Safety population is defined by all phase 1 and phase 2a patients who received at least 1 administration of monalizumab were evaluable for progression-free survival and overall survival efficacy outcomes and for safety. 22 patients were included in the ITT / Safety population.
Arm/Group | ITT / Safety Population
Number analyzed (Participants) | 22
Month | NA [NA to NA] — A PFS median could not be estimated at the time of data cut-off.

6. Secondary Outcome: Overall Survival
Description: The overall survival (OS) is defined as the time from first dose administration until death from any cause. Alive patients were censored at the most recent date they were known to be alive. Subjects with no assessment post-Baseline were censored at the day of the first dose administration.
Time Frame: Up to 24 months.
Population: 22 patients were included in the ITT / Safety population
Measure: Median (95% Confidence Interval); unit: Month
Groups:
- All ITT / Safety Population: The Intent-To-Treat / Safety population is defined by all phase 1 and phase 2a patients who received at least 1 administration of monalizumab were evaluable for progression-free survival and overall survival efficacy outcomes and for safety. 22 patients were included in the ITT / Safety population.
Arm/Group | All ITT / Safety Population
Number analyzed (Participants) | 22
Month | NA [NA to NA] — At the time of data cut-off, all 22 phase 1 and phase 2 patients were alive.

ADVERSE EVENTS:
Time Frame: The occurrences of Adverse Events were recorded from the time of signed informed consent until the end of the patient's participation to the trial (up to 24 months).
Groups:
- 1 mg/kg: During phase 1b, patients received monalizumab, IV, at the dose of 1mg/kg, in combination with ibrutinib 420 mg, orally, once daily.
- 2 mg/kg: During phase 1b and during phase 2a patients received monalizumab, IV, at the dose of 2 mg/kg, in combination with ibrutinib 420 mg, orally, once daily.
- 4 mg/kg: During phase 1b, patients receivde monalizumab, IV, at the dose of 4 mg/kg, in combination with ibrutinib 420 mg, orally, once daily.
Arm/Group | 1 mg/kg | 2 mg/kg | 4 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/15 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/3 | 5/15 | 3/4
Other Adverse Events (participants affected / at risk) | 3/3 | 15/15 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg/kg (N=3) | 2 mg/kg (N=15) | 4 mg/kg (N=4)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 mg/kg (N=3) | 2 mg/kg (N=15) | 4 mg/kg (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (2)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (5) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 9 (15) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 4 (5) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 6 (9) | 2 (4)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 4 (4) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cyst rupture (General disorders) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 4 (4) | 1 (1)
Feeling jittery (General disorders) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 2 (3) | 0 (0)
Mass (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Oedema (General disorders) | 1 (2) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (6) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 2 (5) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 8 (13) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 2 (3) | 0 (0)
Weight increased (Investigations) | 1 (1) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (12) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 7 (8) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 5 (6) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 4 (4) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Onychalgia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (15) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (4) | 7 (20) | 2 (3)

LIMITATIONS AND CAVEATS:
Due to early termination some of the secondary endpoints could not be evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT02557516/SAP_000.pdf
  • Study Protocol (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT02557516/Prot_001.pdf